CLINICAL TRIAL: NCT04803617
Title: The Effect of Pectoralis Muscle Strength on Pulmonary Function in Elderly With Interstitial Lung Disease
Brief Title: Investigation of Pectoralis Muscle Strength in Elderly With Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Habibedurdu (Other)
Responsible Party: Sponsor-Investigator, Habibedurdu, MSc, Giresun University
Organization: Giresun University (Other)
Other Study IDs: Pectoralismajor
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Sarcoidosis, Pulmonary; Geriatric
Keywords: pectoralis muscle strength; lung function test; respiratory muscle strength; horizontal adduction
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Sarcoidosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient's group: geriatric patients with interstitial lung disease
  Interventions: Other: Assessment of pulmonary function and pectoralis muscle strength
- Control group: healthy volunteers selected from the geriatric population
  Interventions: Other: Assessment of pulmonary function and pectoralis muscle strength

INTERVENTIONS:
Other: Assessment of pulmonary function and pectoralis muscle strength — In both groups, forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and FEV1 / FVC ratio were measured with portable spirometer according to the guidelines of the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Maximal inspiratory (MIP) and expiratory pressure (MEP) were evaluated with mouth pressure device as per ATS/ERS guidelines. Sensation of dyspnea was assessed with Modified medical council research scale. Pectoralis muscle strength were measured isometrically using with digital hand held dynamometer.

SUMMARY:
Interstitial lung disease (ILD) is a restrictive lung disease characterized by impaired lung function, exercise limitation and skeletal muscle dysfunction. There is limited data on skeletal muscle function in ILD, most of which are focused on the lower limb muscles. The aim of this study were to evaluated the change of pectoralis muscle strength and relationship of pulmonary function with pectoralis muscle strength.

DETAILED DESCRIPTION:
This study consisted of intervention and control groups. Thirty one patients with ILD were included in the patient's group and 37 healthy volunteers in the control group. All participants were selected from the geriatric population. Demographic and cardiopulmonary physiotherapy assessment of all participants were performed. Lung function test, maximal inspiratory and expiratory pressure and pectoralis muscle strength were measured in participants of both groups. All measurements were performed once.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ILD by a multidisciplinary team according to the 2011 ATS/ERS guidelines for ILD
* Aged 65-85

Exclusion Criteria:

* Uncontrolled/active cardiovascular, metabolic, systemic or cancerous disease
* Significant orthopedic, neurologic or musculoskeletal comorbidity that limited functional independence
* No being able to cooperate
* Refuse to participate in the current study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The patient's group was selected from among the patients who applied to Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital.
  The control group was selected among volunteers invited from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Pectoralis muscle strength test | 15 minute
  The pectoralis muscle strength were measured with handheld dynamometer in supine position. The shoulder joint of participant was positioned at 90º abducted and at 0º internal/external rotation and the elbow joint was flexed at 90º. The other shoulder joint was fixed by the physiotherapist. While the participant performed isometrically horizontal adduction movement, the measurement was performed on the distal part of the upper arm and the contraction was sustained for at least 5 seconds by the participant. The test was performed three times and with 60 seconds rest between tests. The mean of the best value on both sides was recorded.

SECONDARY OUTCOMES:
FEV1 | 5 minute
  FEV1 value was measured with portable spirometer according to ATS/ ERS guidelines for pulmonary function test. Results of the measurements were recorded as percentanges of predicted values.
FVC | 5 minute
  FVC value was measured with portable spirometer according to ATS/ ERS guidelines for pulmonary function test. Results of the measurements were recorded as percentanges of predicted values.
FEV1/FVC | 5 minute
  The ratio of FEV1/FVC was calculated by measuring device according to measured FEV1 and FVC values
Respiratory muscle strength test | 15 minute
  Maximal mouth pressures were measured to evaluate respiratory muscle strength. The test was performed with mouth pressure device in sitting position. Participants breathed through a flanged mouthpiece inside the lips at near residual volume for the MIP value and near total lung capacity for MEP value . The maximum effort was sustained for at least one second. The test was repeated at least 3 times until no more than 10% difference was present between highest and previous measurements . The higest value and percentage value of predicted highest value were recorded
Dyspnea assessment | 3 minute
  Modified Medical Council Research Dyspnea scale were used to assess sensation of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Habibe DURDU, MSc, Principal Investigator — Giresun University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sets collected and analyzed during this study could be provided from corresponding author upon reasonable request

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Result] Hirano M, Katoh M, Kawaguchi S, Uemura T. Intrarater reliabilities of shoulder joint horizontal adductor muscle strength measurements using a handheld dynamometer for geriatric and stroke patients. J Phys Ther Sci. 2016 Jan;28(1):51-5. doi: 10.1589/jpts.28.51. Epub 2016 Jan 30. PMID 26957727
- [Result] Panagiotou M, Polychronopoulos V, Strange C. Respiratory and lower limb muscle function in interstitial lung disease. Chron Respir Dis. 2016 May;13(2):162-72. doi: 10.1177/1479972315626014. Epub 2016 Jan 14. PMID 26768011
- [Result] Hanada M, Sakamoto N, Ishimatsu Y, Kakugawa T, Obase Y, Kozu R, Senjyu H, Izumikawa K, Mukae H, Kohno S. Effect of long-term treatment with corticosteroids on skeletal muscle strength, functional exercise capacity and health status in patients with interstitial lung disease. Respirology. 2016 Aug;21(6):1088-93. doi: 10.1111/resp.12807. Epub 2016 May 13. PMID 27173103
- [Derived] Durdu H, Yurdalan SU, Ozmen I. Clinical significance of pectoralis muscle strength in elderly patients with idiopathic pulmonary fibrosis. Sarcoidosis Vasc Diffuse Lung Dis. 2022;39(1):e2022009. doi: 10.36141/svdld.v39i1.12094. Epub 2022 Mar 31. PMID 35494168